CLINICAL TRIAL: NCT06176404
Title: Stellate Ganglion Block in Cerebral Small Vessel Disease Patients With Dysphagia and Cognitive Impairment
Brief Title: Stellate Ganglion Block in Patients With Cerebral Small Vessel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeng Changhao (Other)
Responsible Party: Sponsor-Investigator, Zeng Changhao, Research Director, People's Hospital of Zhengzhou University
Organization: People's Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NXXG-SGB-jiu
Record Dates: First submitted 2023-12-11; First posted 2023-12-19 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Dysphagia; Cerebral Small Vessel Diseases; Cognitive Impairment
MeSH Terms: conditions — Deglutition Disorders; Cerebral Small Vessel Diseases; Cognitive Dysfunction | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The comparison group (Active Comparator): The study lasted 20d for each patient. During the treatment, All the participants were provided with the rehabilitation therapy, which included routine rehabilitation, cognitive training, swallowing function training and nutrition support.
  Particularly, due to dysphagia, the patients enrolled might face difficulty in eating. For patients who were able to finish intake via mouth by compensatory means, the consistency, type, and size of food bolus was arranged. For those who cannot acquire sufficient nutrition through oral intake, the nasogastric tube feeding (NGT) was provided.
  Interventions: Behavioral: Rehabilitation therapy
- The observation group (Experimental): The study lasted 20d for each patient. During the treatment, All the participants were provided with the rehabilitation therapy, which included routine rehabilitation, cognitive training, swallowing function training and nutrition support.
  Particularly, due to dysphagia, the patients enrolled might face difficulty in eating. For patients who were able to finish intake via mouth by compensatory means, the consistency, type, and size of food bolus was arranged. For those who cannot acquire sufficient nutrition through oral intake, the nasogastric tube feeding (NGT) was provided.
  Based on the invention above, the patients in the observation group were provided with SGB, using 1.5ml of 2% Lidocaine hydrochloride (1ml: 0.5mg) and 500ug of Vitamin B12 (1ml: 0.5g).
  Interventions: Drug: Stellate ganglion block; Behavioral: Rehabilitation therapy

INTERVENTIONS:
Drug: Stellate ganglion block — Based on the invention above, the patients in the observation group were provided with SGB, using 1.5ml of 2% Lidocaine hydrochloride (1ml: 0.5mg) and 500ug of Vitamin B12 (1ml: 0.5g). The percutaneous approach via the paratracheal route was used for SGB. The operator stood on the side of the block, instructed the patient to lie supine with a thin pillow placed below the shoulders, and tilted the head 45° towards the blocked side, fully exposing the neck. Then, routine disinfection of the neck skin was performed. The puncture site was located 2.5 cm above the sternoclavicular joint and 1.5 cm lateral to the midline of the neck.
  Other Names: SGB
  Arms: The observation group
Behavioral: Rehabilitation therapy — The study lasted 20d for each patient. During the treatment, All the participants were provided with the rehabilitation therapy, which included routine rehabilitation, cognitive training, swallowing function training and nutrition support.
  Particularly, due to dysphagia, the patients enrolled might face difficulty in eating. For patients who were able to finish intake via mouth by compensatory means, the consistency, type, and size of food bolus was arranged. For those who cannot acquire sufficient nutrition through oral intake, the nasogastric tube feeding (NGT) was provided.
  Other Names: Rehabilitation Treatment

SUMMARY:
A prospective study was conducted on 84 CSVD patients with dysphagia and cognitive impairment. They were divided into the comparison group and observation group evenly. All the patients were provided with routine therapy, while the patients in the observation group were given SGB. The swallowing function, cognitive function and activities of daily living of the two groups of patients before and after treatment were evaluated by Penetration-Aspiration Scale, Mini-mental state examination and modified Barthel index.

DETAILED DESCRIPTION:
In order to observe the effect of stellate ganglion block (SGB) on swallowing function, cognitive function and activities of daily living in patients with cerebral small vessel disease (CSVD), A prospective study was conducted on 84 CSVD patients with dysphagia and cognitive impairment. They were divided into the comparison group and observation group evenly. All the patients were provided with routine therapy, while the patients in the observation group were given SGB. The swallowing function, cognitive function and activities of daily living of the two groups of patients before and after treatment were evaluated by Penetration-Aspiration Scale, Mini-mental state examination and modified Barthel index.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years.
* Meeting the diagnostic criteria for cerebral small vessel disease Imaging proposed in 2013 by the international cerebral small vessel disease Expert Group, and the "Consensus on Diagnosis and Treatment of Cerebral Small Vessel Disease in China" in 2017.
* Dysphagia confirmed by Videofluoroscopic Swallowing Study
* Mini-Mental State Examination (MMSE)<27, indicating the existence of cognitive impairment.
* No history of prior stroke.
* Stable vital signs.

Exclusion Criteria:

* Dysphagia that might be caused by other diseases that might cause dysphagia, such as head and neck tumors, traumatic brain injury, myasthenia gravis, etc.
* Cognitive impairment that might be caused by other diseases, such as Alzheimer's disease, Parkinson's disease, brain injury, etc.
* Neurological blockade contraindications such as bleeding tendency, blocked site infection.
* MMSE<10, or unable to successfully finish the assessment of this study (Patients with severe mental illness or intellectual disability might have difficulty to cooperate with the assessment).
* Complicated with severe liver and kidney failure, tumors, or hematological disorders.
* Simultaneously in need to undergo other therapy that might affect the outcomes of this study.
* Pregnant or nursing females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Penetration-Aspiration Scale | day 1 and day 20
  On the day 1 and day 20, Penetration-Aspiration Scale was used to assess dysphagia under Videofluoroscopic Swallowing Study, primarily evaluating the extent to which fluid food entered the airway and caused penetration or aspiration during the swallowing process. As the level increased, the severity of dysphagia also increased.

SECONDARY OUTCOMES:
Modified Barthel Index | day 1 and day 20
  On the day 1 and day 20, the activities of daily living of patients were assessed using the modified Barthel Index . The scale included 10 items such as feeding, bathing, walking, dressing. Each item was rated on a 4-point scale based on the level of assistance required, with a total score of 100 points. There was a positive correlation between activities of daily living and the final score.
Mini-Mental State Examination | day 1 and day 20
  On the day 1 and day 20, the cognitive function of patients was assessed using the Mini-Mental State Examination (MMSE). The MMSE evaluated five aspects, including orientation, memory, attention and calculation abilities, recall ability, and language skills, with a total score of 30 points. A MMSE score of less than 27 indicated cognitive impairment, with scores ≤9 indicating severe impairment, 10-20 indicating moderate impairment, and 21-26 indicating mild impairment.
Swallowing duration | day 1 and day 20
  The time duration that the patient swallowed the contrast agent under Videofluoroscopic Swallowing Study the was recorded.Unit: seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Principal Investigator — Site Coordinator of United Medical Group located in Miami
Locations (1):
- Zhen Da No.1 Fushu Hos., Huabei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zeng H, Zhao W, Fang L, Pan H, Huang S, Zeng X. Effect of Stellate Ganglion Block on Dysphagia and Cognitive Impairment in Cerebral Small Vessel Disease: A Randomized Controlled Study. J Speech Lang Hear Res. 2024 Oct 8;67(10):3660-3672. doi: 10.1044/2024_JSLHR-24-00145. Epub 2024 Sep 13. PMID 39270205